CLINICAL TRIAL: NCT03798496
Title: Role of the Interosseous Membrane and TFCC in DRUJ Stability in Galeazzi´s Fracture: Anatomical and Biomechanical Study
Brief Title: Anatomical and Biomechanical Study About Stability in Galeazzi´s Fracture
Acronym: Galeazzi
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-GAL-2018-75
Record Dates: First submitted 2018-12-19; First posted 2019-01-10 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Galeazzi's Fracture
MeSH Terms: conditions — Radius Fractures | interventions — Open Fracture Reduction; Fracture Fixation, Internal; Bone Wires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Open reduction and internal fixation — Open reduction of the Galeazzi fracture dislocation with a plate.
  Other Names: DRUJ reduction with Kirschner wire

SUMMARY:
Most Galeazzi fractures can be treated adequately with open reduction and internal fixation (ORIF) of the radius alone, but some will remain unstable at the DRUJ and require repair of the TFCC.The purpose of this anatomical and biomechanical study was to define and measure DRUJ dislocation, displacement and instability associated with the sequential sectioning of the different bands in the interosseous membrane (IOM) and TFCC in the simulation of a Galeazzi fracture.

DETAILED DESCRIPTION:
Instability of the DRUJ is a common clinical problem associated with Galeazzi fracture. Stability of the DRUJ is primarily provided by both the bony anatomy of the sigmoid notch of the radius and ulnar head and the soft tissues surrounding the joint. The interosseous membrane plays an important role in DRUJ stability but the TFCC is the major soft tissue stabilizer of the DRUJ. The Central Band works as a restraint on the radius from proximal migration in cooperation with the radial head and the TFCC and also works as a load transmitter between the radius and ulnar to redistribute load. Some investigators suggested that the distal membranous portion and DOB stabilizes the DRUJ when TFCC is disrupted. Watanabe et al. (2005) insisted on the importance of DOB, which constrained volar and dorsal instability of the radius at the DRUJ in all forearm rotation positions. The purpose of this anatomical and biomechanical study was to define and measure DRUJ dislocation in the simulation of a Galeazzi fracture.

ELIGIBILITY:
Inclusion Criteria:

Adults patients(18-85 years old) with Galeazzi fracture-dislocation treated with open reduction and internal fixation (ORIF).

Exclusion Criteria:

* Children
* Other types of forearms fractures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anatomical and biomechanical study: Twelve specimens from the Human Anatomy Department.
  Clinical study: Review of reports (X-rays) about patients with Galeazzi fracture-dislocation treated with ORIF.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Displacement in distal radius fracture | 12 months
  The investigators will mesure the degree of displacement (mm) in a simulate distal radius fracture with a biomechanical device named Medmesin with a especific computer software that applies newtons (from 0 to 100N) in the radius in each especimen.
Stability in the DRU joint | 12 months
  Dislocation of the ulnar in the wrist. In the retrospective clinical reports the investigators evaluate the x-rays before and after the surgery and the radioulnar ratio in the CT scan (congruency method, Mino criteria and the epicenter method).

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Lamas, Ph D, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
After the results were obtained we send the results to the statistical department to correlate the outcomes.

REFERENCES:
- [Background] Farr LD, Werner FW, McGrattan ML, Zwerling SR, Harley BJ. Anatomy and biomechanics of the forearm interosseous membrane. J Hand Surg Am. 2015 Jun;40(6):1145-51.e2. doi: 10.1016/j.jhsa.2014.12.025. Epub 2015 Feb 20. PMID 25703865
- [Background] Kitamura T, Moritomo H, Arimitsu S, Berglund LJ, Zhao KD, An KN, Rizzo M. The biomechanical effect of the distal interosseous membrane on distal radioulnar joint stability: a preliminary anatomic study. J Hand Surg Am. 2011 Oct;36(10):1626-30. doi: 10.1016/j.jhsa.2011.07.016. Epub 2011 Aug 26. PMID 21872404
- [Background] Loeffler BJ, Green JB, Zelouf DS. Forearm instability. J Hand Surg Am. 2014 Jan;39(1):156-67. doi: 10.1016/j.jhsa.2013.07.010. Epub 2013 Dec 6. PMID 24315636
- [Background] Moritomo H. The distal interosseous membrane: current concepts in wrist anatomy and biomechanics. J Hand Surg Am. 2012 Jul;37(7):1501-7. doi: 10.1016/j.jhsa.2012.04.037. PMID 22721462
- [Background] Noda K, Goto A, Murase T, Sugamoto K, Yoshikawa H, Moritomo H. Interosseous membrane of the forearm: an anatomical study of ligament attachment locations. J Hand Surg Am. 2009 Mar;34(3):415-22. doi: 10.1016/j.jhsa.2008.10.025. Epub 2009 Feb 11. PMID 19211201
- [Background] Petersen MS, Adams BD. Biomechanical evaluation of distal radioulnar reconstructions. J Hand Surg Am. 1993 Mar;18(2):328-34. doi: 10.1016/0363-5023(93)90370-I. PMID 8463602
- [Background] Riggenbach MD, Conrad BP, Wright TW, Dell PC. Distal oblique bundle reconstruction and distal radioulnar joint instability. J Wrist Surg. 2013 Nov;2(4):330-6. doi: 10.1055/s-0033-1358546. PMID 24436838
- [Background] Riggenbach MD, Wright TW, Dell PC. Reconstruction of the Distal Oblique Bundle of the Interosseous Membrane: A Technique to Restore Distal Radioulnar Joint Stability. J Hand Surg Am. 2015 Nov;40(11):2279-82. doi: 10.1016/j.jhsa.2015.08.019. PMID 26518322
- [Background] Werner FW, LeVasseur MR, Harley BJ, Anderson A. Role of the Interosseous Membrane in Preventing Distal Radioulnar Gapping. J Wrist Surg. 2017 May;6(2):97-101. doi: 10.1055/s-0036-1584545. Epub 2016 Jun 20. PMID 28428910
- [Background] Werner FW, Taormina JL, Sutton LG, Harley BJ. Structural properties of 6 forearm ligaments. J Hand Surg Am. 2011 Dec;36(12):1981-7. doi: 10.1016/j.jhsa.2011.09.026. Epub 2011 Nov 17. PMID 22100813